CLINICAL TRIAL: NCT02013960
Title: Comparison Between Sublingual Misoprostol vs. Sublingual Misoprostol and Laminaria For Second Trimester Termination of Pregnancy
Brief Title: Misoprostol vs. Sublingual Misoprostol and Laminaria For Second Trimester Termination of Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Awad Nibal MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0099-13-RMB CTIL
Record Dates: First submitted 2013-09-16; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Other Abortion
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laminaria (Experimental): cytotec and laminaria
  Interventions: Drug: Cytotec
- Cytotec (Active Comparator): Cytotec only
  Interventions: Drug: Cytotec

INTERVENTIONS:
Drug: Cytotec — Cytotec medication compared with cytotec and laminaria
  Other Names: Misorpristol vs. Misopristol and laimnria

SUMMARY:
1. Comparison between the duration of time from the beginning of cervical preparation until abortion, between sublingual misoprostol and the combination of sublingual misoprostol with laminaria for second trimester medical termination of pregnancy (TOP).
2. Comparison between the adverse event rate following Sublingual misoprostol only vs. Sublingual misoprostol and laminaria given for pregnancy termination.
3. Comparison between the levels of satisfaction rate of women who underwent pregnancy termination with sublingual misoprostol vs. sublingual misoprostol with laminaria.

DETAILED DESCRIPTION:
A prospective randomized control trial; 50 women undergoing pregnancy termination in the second trimester (14-28 weeks)in each group.

Following receiving an ethical approval by the local institutional review board (IRB), committee, consecutively all women in between 14 weeks to 28 weeks; that have a reason for termination of pregnancy like: intrauterine fetal death or medical or genetic indications for termination of pregnancy or socioeconomic termination of pregnancy will be offered to take part in the study. If eligible according to the inclusion and exclusion criteria, women will be asked to sign a consent form.

All participants will undergo blood exams (CBC, Prothrombin time, Partial thromboplastin time , and BLOOD TYPING) and ultrasound exam for Confirmation of diagnosis as routinely indicated for missed abortion at our department

ELIGIBILITY:
Inclusion Criteria:

Second trimester pregnancy No evidence of chorioamnionitis

Exclusion Criteria:

Allergy to misoprostol. Evidence for infection. Asthma

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Duration of time until pregnancy termination | Average time 12 hours
  From the time of receiving the treatment until complete abortion

CONTACTS AND LOCATIONS:
Overall Officials: Nibal Awad, MD, Study Chair — Rambam Health Care Campus
Locations (1):
- Rambam Health Campus, Haifa, Israel